CLINICAL TRIAL: NCT06404918
Title: Comparison Between Preemptive Erector Spinae Plane Block Versus Serratus Anterior Plane Block on Postoperative Analgesia for Patients Undergoing Modified Radical Mastectomy: A Randomized Clinical Trial
Brief Title: Preemptive Erector Spinae Plane Block Versus Serratus Anterior Plane Block in MRM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ramy Mousa, Professor, Benha University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RC 23-11-2023
Record Dates: First submitted 2024-05-01; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-04

CONDITIONS: Modified Radical Mastectomy
Keywords: Erector Spinae Plane Block; Serratus Anterior Plane Block

STUDY DESIGN:
Intervention Model Description: Group I (35 patients): patients received US ESPB and group II (35 patients): patients received USAPB.
Who Masked: Participant, Care Provider
Masking Description: The patients and Care Provider in this trial were blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector spinae plane group (Experimental): The patients were placed in lateral decubitus position with the operation site up. The probe was placed vertically 3 cm lateral to the T5 spinous process, and the transverse process was identified as an oval hyperechoic sonographic structure. The needle was introduced in an in-plane fashion until the tip lay deep in the erector spinae muscle. 0.5 mL of normal saline was injected to confirm the correct needle tip position by visualizing the spread under the erector spinae muscle. A total of 0.4 mL kg-1 of 0.25% bupivacaine was injected. between the erector spinae muscle and transverse process.
  Interventions: Procedure: Erector spinae plane group
- Serratus anterior plane group (Experimental): Serratus anterior plane block was administered to patient in the supine position with ipsilateral arm abducted to 90°. Under aseptic precautions, linear probe was placed over the midclavicular region in the sagittal plane. Ribs were counted inferiorly and laterally until the fifth rib was identified in midaxillary line. Latissimus dorsi, teres major, and serratus anterior muscles were identified overlying the fifth rib. The intended puncture site was infiltrated with 2 mL of 2% lignocaine, and using ultrasound-guided in-plane approach, the needle was introduced in caudal to cranial direction until the tip was placed between the serratus anterior muscle and external intercostal muscle.
  Interventions: Procedure: Serratus anterior plane group

INTERVENTIONS:
Procedure: Erector spinae plane group — The patients were placed in lateral decubitus position with the operation site up. The probe was placed vertically 3 cm lateral to the T5 spinous process, and the transverse process was identified as an oval hyperechoic sonographic structure. The needle was introduced in an in-plane fashion until the tip lay deep in the erector spinae muscle. 0.5 mL of normal saline was injected to confirm the correct needle tip position by visualizing the spread under the erector spinae muscle. A total of 0.4 mL kg-1 of 0.25% bupivacaine was injected. between the erector spinae muscle and transverse process.
  Other Names: US ESPB group
  Arms: Erector spinae plane group
Procedure: Serratus anterior plane group — Serratus anterior plane block was administered to patient in the supine position with ipsilateral arm abducted to 90°. Under aseptic precautions, linear probe was placed over the midclavicular region in the sagittal plane. Ribs were counted inferiorly and laterally until the fifth rib was identified in midaxillary line. Latissimus dorsi, teres major, and serratus anterior muscles were identified overlying the fifth rib. The intended puncture site was infiltrated with 2 mL of 2% lignocaine, and using ultrasound-guided in-plane approach, the needle was introduced in caudal to cranial direction until the tip was placed between the serratus anterior muscle and external intercostal muscle.
  Other Names: USAPB group
  Arms: Serratus anterior plane group

SUMMARY:
Modified radical mastectomy (MRM) is one of the most performed surgeries for breast cancer. MRM is associated with significant pain during the immediate postoperative period.

DETAILED DESCRIPTION:
Modified radical mastectomy (MRM) is one of the most performed surgeries for breast cancer. MRM is associated with significant pain during the immediate postoperative period.

Inadequate pain management has both psychological and physiological repercussions.

Various local or regional nerve blocks like thoracic epidural, interscalene brachial plexus, paravertebral, pectoral nerve blocks, and erector spinae plane blocks are performed in MRM to provide analgesia.

Ultrasound-guided Erector spinae plane block (USG-ESPB) is one of the novel and effective regional techniques where local anaesthetic is deposited deep into the erector spinae muscle, blocking the ventral and dorsal rami of multiple spinal nerves, and is technically simple, with fewer hemodynamic side effects and with minimal complications

ELIGIBILITY:
Inclusion Criteria:

* female patients
* aged from 18 to 70 years
* with a body mass index ≤ 30 kg/ m2
* American Society of Anesthesiologists (ASA) physical status I-II,
* who were scheduled for MRM for breast cancer

Exclusion Criteria:

* history of drug allergy,
* psychiatric illness, substance abuse,
* severe cardiovascular or respiratory disease,
* any pre-existing liver disease, metabolic or neurological syndrome, c

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 70 (Actual)
Dates: Start 2023-01-22 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2024-04-03 (Actual)

PRIMARY OUTCOMES:
time of the first rescue analgesic dose | 24 hours postoperatively
  The time when the first dose of rescue analgesia was administered at the recovery room,

SECONDARY OUTCOMES:
Heart rate changes | 15 minutes after performing the block, and then every 30 minutes intraoperatively till the end of surgery, then postoperatively at 1hour and 2 hours, 4hours, 8hours, 12hours, 18hours, 24hours postoperatively.
  Heart rate (HR) was recorded immediately before induction of anaesthesia, 1
Mean arterial pressure changes | 15 minutes after performing the block, and then every 30 minutes intraoperatively till the end of surgery, then postoperatively at 1hour and 2 hours, 4hours, 8hours, 12hours, 18hours, 24hours postoperatively.
  Mean arterial pressure

CONTACTS AND LOCATIONS:
Overall Officials: Ramy Saleh, MD, Principal Investigator — Anesthesia and surgical ICU department, Faculty of Medicine, Benha University, Egypt
Locations (1):
- Benha University, Banhā, Egypt

IPD SHARING:
Plan to Share IPD: No